CLINICAL TRIAL: NCT07243041
Title: A Prospective Study Exploring Factors Affecting ICU Transitions and Handling of Code Status - Insights Into Physician and Family Communication in a Muslim Patient Population
Brief Title: Code Status Discussions in Muslim ICU Patients: Insights Into Physician-Family Communication
Acronym: FAITH-ICU
Status: Recruiting | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Imran Khalid, Consultant, King Faisal Specialist Hospital & Research Center
Other Study IDs: 2251305
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: End of Life Care; Muslim; Decision Making ,Shared
Keywords: goals of care; do not attempt resuscitation; ICU; Shared Decision-Making; Family Communication; Muslim Healthcare Context; Cultural Factors; palliative care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU DNAR Discussion Episodes: Adult ICU patients with DNAR discussions during the study period. Observational study; no interventions. Physicians complete post-discussion questionnaires, and limited retrospective EMR data are collected to examine factors influencing DNAR decision outcomes, including final code status

SUMMARY:
This observational study aims to explore the real-time experiences, perceptions, and challenges faced by intensive care unit (ICU) physicians during goals-of-care discussions-specifically Do Not Attempt Resuscitation (DNAR) and end-of-life decision-making conversations-with families of critically ill patients in a Muslim-majority healthcare setting.

The study seeks to identify factors that influence whether a DNAR decision is reached after physician-family discussions, and how physician experience, family dynamics, religious perspectives, and institutional support affect communication outcomes and care transitions.

Participants will include ICU physicians (residents, fellows, and consultants) who routinely conduct DNAR discussions as part of clinical care. After each discussion, physicians will complete a brief structured questionnaire about their perceptions of the interaction, family emotions, and decision outcomes. These responses will be anonymously linked to limited, de-identified patient-level data (e.g., diagnosis, ICU course, and outcome) extracted retrospectively from the electronic medical record.

No patients or family members will be contacted directly. Data collection will occur prospectively over two years at King Faisal Specialist Hospital & Research Centre-Jeddah.

Findings from this study are expected to provide culturally grounded insights that inform physician training, enhance family-centered communication, and guide policy development for DNAR and end-of-life discussions in Muslim-majority intensive care units.

DETAILED DESCRIPTION:
Background:

This prospective observational study investigates the real-time experiences, perceptions, and challenges faced by ICU physicians when discussing code status decisions, specifically Do Not Attempt Resuscitation (DNAR), with families of critically ill adult patients in a Muslim-majority healthcare context. It aims to identify clinical, cultural, religious, and institutional factors influencing DNAR discussions, addressing a gap in understanding the interpersonal and theological dynamics that shape decision-making in end-of-life care. Findings will inform culturally sensitive communication practices, policy development, and physician training.

Study Design and Setting:

Prospective, mixed-methods observational study over 24 months (November 2025 - October 2027). Conducted in adult ICUs at King Faisal Specialist Hospital & Research Centre (KFSH&RC), Jeddah. Integrates real-time physician survey data immediately after DNAR discussions with retrospective EMR extraction of patient-level variables. A subsequent qualitative phase with physician interviews will contextualize quantitative findings. No patients or families are directly contacted.

Definitions of DNAR:

Full Resuscitation: Eligible for all life-sustaining interventions (CPR, intubation, mechanical ventilation, vasopressors).

Ward-Level DNAR: Primarily comfort-focused; prohibits CPR/intubation but allows non-invasive supportive care; home ventilator patients may continue care; ICU transfer allowed per order.

ICU-Level DNAR: Allows withholding or withdrawal of life-sustaining interventions within predefined ceilings:

1. Without interventions: Comfort measures only, no invasive procedures.
2. With interventions: Selected invasive therapies (vasopressors, RRT, non-invasive ventilation, cardioversion) allowed, but no ACLS/chest compressions/intubation if not already intubated.

Therapy may be capped at a defined level; full-code patients may convert to ICU-level DNAR during ICU stay.

Study Population:

ICU physicians (residents, fellows, assistant consultants, consultants) conducting DNAR discussions with adult patients' families. Participation is voluntary; physicians who decline or discuss patients <18 years old are excluded.

Outcomes:

Primary: Final code status immediately post-discussion (DNAR [with/without limited interventions] vs. Full Code).

Secondary: Timing and emotional tone of discussions, family conflict/resolution, institutional support, physician experience/confidence, and quality of end-of-life care using ICU-adapted Aggressive Care and Comfort-Oriented (Palliation) Composites in the final 24 hours of life.

Analysis:

Target 320-500 completed DNAR discussion episodes, accounting for clustering by physician.

Primary analysis via mixed-effects logistic regression with up to 11 pre-specified predictors (physician, family, and clinical/timing factors).

Secondary analyses explore associations with ICU course, timing, composite indices, and comparisons with patients without DNAR discussions.

Sensitivity and subgroup analyses include early vs late discussions (≤72h vs >72h) and cancer vs non-cancer diagnoses.

If fewer than 320 completed DNAR discussions are collected within the planned study period, the study duration may be extended to achieve the minimum sample size required for reliable multivariable analysis.

Data Protection and Ethics:

Each questionnaire linked to de-identified EMR data via unique study ID; master linkage file securely stored and encrypted. Physician participation implies consent; retrospective EMR review conducted under a waiver of consent per institutional and international guidelines.

Expected Outcomes:

The study will generate empirical, culturally grounded insights into DNAR discussions in Muslim-majority ICUs, clarifying how physician experience, family dynamics, and religious or institutional context shape communication. Results will guide physician training, policy frameworks, and family-centered, ethically sound end-of-life care practices.

ELIGIBILITY:
Inclusion Criteria:

* ICU physicians (residents, fellows, assistant consultants, or consultants) involved in direct patient care
* ICU physicians who conduct code status or Do Not Attempt Resuscitation (DNAR) discussions with patients' families during ICU admission
* Willingness of ICU physicians to participate voluntarily by completing a post-goals-of-care discussion questionnaire
* Adult patients (≥18 years) admitted to the ICU during the study period for whom a code status discussion occurred

Exclusion Criteria:

* ICU physicians who decline participation
* Code status discussions involving patients younger than 18 years of age
* Discussions in which the physician was not directly involved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients (≥18 years) for whom a code status discussion regarding Do Not Attempt Resuscitation (DNAR) occurs during the study period (November 2025 to October 2027). Participating ICU physicians will complete a structured post-discussion questionnaire. Limited retrospective patient data will be extracted from the electronic medical record to characterize clinical context, ICU course, and outcomes. The study includes all eligible ICU physicians involved in these discussions who consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Do Not Attempt Resuscitation (DNAR) Status After Goals-of-Care Discussion | After each DNAR discussion
  Final resuscitation status immediately following each goals-of-care discussion, categorized as Do Not Attempt Resuscitation (DNAR, including DNAR with or without limited interventions) versus Full Code.
  The outcome will be analyzed as a binary variable representing whether DNAR status was established following the discussion.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Khalid, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the study team. All data will remain confidential and stored securely according to institutional policies

REFERENCES:
- [Background] Wachterman MW, Pilver C, Smith D, Ersek M, Lipsitz SR, Keating NL. Quality of End-of-Life Care Provided to Patients With Different Serious Illnesses. JAMA Intern Med. 2016 Aug 1;176(8):1095-102. doi: 10.1001/jamainternmed.2016.1200. PMID 27367547
- [Background] Teno JM, Gozalo PL, Bynum JP, Leland NE, Miller SC, Morden NE, Scupp T, Goodman DC, Mor V. Change in end-of-life care for Medicare beneficiaries: site of death, place of care, and health care transitions in 2000, 2005, and 2009. JAMA. 2013 Feb 6;309(5):470-7. doi: 10.1001/jama.2012.207624. PMID 23385273
- [Background] Hui D, Kim SH, Roquemore J, Dev R, Chisholm G, Bruera E. Impact of timing and setting of palliative care referral on quality of end-of-life care in cancer patients. Cancer. 2014 Jun 1;120(11):1743-9. doi: 10.1002/cncr.28628. PMID 24967463
- [Background] Clarke EB, Curtis JR, Luce JM, Levy M, Danis M, Nelson J, Solomon MZ; Robert Wood Johnson Foundation Critical Care End-Of-Life Peer Workgroup Members. Quality indicators for end-of-life care in the intensive care unit. Crit Care Med. 2003 Sep;31(9):2255-62. doi: 10.1097/01.CCM.0000084849.96385.85. PMID 14501954
- [Background] Alao DO, Abraham S, Dababneh E, Roby R, Farid M, Mohammed N, Rojas-Perilla N, Cevik AA. Do-not-attempt-resuscitation decision making: physicians' recommendations differ from the GO-FAR score predictions. Int J Emerg Med. 2024 Jul 11;17(1):86. doi: 10.1186/s12245-024-00669-3. PMID 38992598
- [Background] Padela AI, Zaganjor H. Relationships between Islamic religiosity and attitude toward deceased organ donation among American Muslims: a pilot study. Transplantation. 2014 Jun 27;97(12):1292-9. doi: 10.1097/01.TP.0000441874.43007.81. PMID 24646775
- [Background] Padela AI, Zaidi D. The Islamic tradition and health inequities: A preliminary conceptual model based on a systematic literature review of Muslim health-care disparities. Avicenna J Med. 2018 Jan-Mar;8(1):1-13. doi: 10.4103/ajm.AJM_134_17. PMID 29404267
- [Background] Baykara N, Utku T, Alparslan V, Arslantas MK, Ersoy N. Factors affecting the attitudes and opinions of ICU physicians regarding end-of-life decisions for their patients and themselves: A survey study from Turkey. PLoS One. 2020 May 20;15(5):e0232743. doi: 10.1371/journal.pone.0232743. eCollection 2020. PMID 32433670
- [Background] ur Rahman M, Abuhasna S, Abu-Zidan FM. Care of terminally-ill patients: an opinion survey among critical care healthcare providers in the Middle East. Afr Health Sci. 2013 Dec;13(4):893-8. doi: 10.4314/ahs.v13i4.5. PMID 24940309
- [Background] Saeed F, Kousar N, Aleem S, Khawaja O, Javaid A, Siddiqui MF, Holley JL. End-of-life care beliefs among Muslim physicians. Am J Hosp Palliat Care. 2015 Jun;32(4):388-92. doi: 10.1177/1049909114522687. Epub 2014 Feb 13. PMID 24526765
- [Background] Khalid I, Imran M, Yamani RM, Imran M, Akhtar MA, Khalid TJ. Comparison of Clinical Characteristics and End-of-Life Care Between COVID-19 and Non-COVID-19 Muslim Patients During the 2020 Pandemic. Am J Hosp Palliat Care. 2021 Sep;38(9):1159-1164. doi: 10.1177/10499091211018657. Epub 2021 May 27. PMID 34039050
- [Background] Gouda A, Al-Jabbary A, Fong L. Compliance with DNR policy in a tertiary care center in Saudi Arabia. Intensive Care Med. 2010 Dec;36(12):2149-53. doi: 10.1007/s00134-010-1985-3. Epub 2010 Sep 14. PMID 20838763
- [Background] Rahman MU, Arabi Y, Adhami NA, Parker B, Al-Shimemeri A. The practice of do-not-resuscitate orders in the Kingdom of Saudi Arabia. The experience of a tertiary care center. Saudi Med J. 2004 Sep;25(9):1278-9. No abstract available. PMID 15448786
- [Background] AbuYahya O, Abuhammad S, Hamoudi B, Reuben R, Yaqub M. The do not resuscitate order (DNR) from the perspective of oncology nurses: A study in Saudi Arabia. Int J Clin Pract. 2021 Aug;75(8):e14331. doi: 10.1111/ijcp.14331. Epub 2021 May 17. PMID 33960067
- [Background] Sarhill N, LeGrand S, Islambouli R, Davis MP, Walsh D. The terminally ill Muslim: death and dying from the Muslim perspective. Am J Hosp Palliat Care. 2001 Jul-Aug;18(4):251-5. doi: 10.1177/104990910101800409. PMID 11467099
- [Background] Hamouda MA, Emanuel LL, Padela AI. Empathy and Attending to Patient Religion/Spirituality: Findings from a National Survey of Muslim Physicians. J Health Care Chaplain. 2021 Apr-Jun;27(2):84-104. doi: 10.1080/08854726.2019.1618063. Epub 2019 Jun 10. PMID 31179903